CLINICAL TRIAL: NCT03370029
Title: Comparison of Respiratory Muscle Strength, Exercise Capacity and Physical Activity Levels in Children With Primary Ciliary Dyskinesia and Healthy Controls
Brief Title: Respiratory Muscle Strength, Exercise Capacity and Physical Activity Levels in Children Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: Gazi University5
Record Dates: First submitted 2017-11-10; First posted 2017-12-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Exercise capacity; Respiratory muscle strength; Physical inactivity; Quality of life
MeSH Terms: conditions — Ciliary Motility Disorders; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary ciliary dyskinesia patients: Primary ciliary dyskinesia patients will be included in study. Inclusion and exclusion criteria were considered.
- Healthy individuals: Those without diagnosed chronic disease will be included in study. Inclusion and exclusion criteria were considered.

SUMMARY:
Primary ciliary dyskinesia is an autosomal recessive disorder characterized by abnormal ciliary movement and disrupted mucociliary clearance. In uncleaned airways, microorganisms and respiratory irritants cause inflammation and infection. Permanent rhinitis and chronic sputum cough are typical features in primary ciliary dyskinesia patients. Primary ciliary dyskinesia is a disease that threatens lung function from pre-school age. One of the main causes of respiratory muscle weakness in chronic lung diseases diseases is worsening of lung function. Such a weakness causes alveolar hypoventilation, microatelectasis, reduction of the cough strength .The cough strength is important for airway cleaning.

Exercise capacity is affected in chronic lung diseases. Assessment of exercise capacity in chronic lung diseases is prognostically important. Reduced exercise capacity and pulmonary function in PCD cause decrease in physical activity level. PCD patients have low quality of life and early recognition has been found to affect the quality of life positively. Children with chronic illness have higher level of depression than healthy children.

In literature, no study investigated respiratory muscle strength, exercise capacity and physical activity PCD patients. Therefore, the investigators aimed to compare aforementioned outcomes in PCD patients and healthy controls.

DETAILED DESCRIPTION:
According to sample size calculation 26 diagnosed primary ciliary dyskinesia patients and 26 healthy individuals will be included. Respiratory muscle strength, anaerobic and aerobic exercise capacity, physical activity, pulmonary functions, peripheral muscle strength, cough strength, respiratory muscle endurance, activity dyspnea perception, quality of life and depression will be evaluated. Primary outcome measurements are respiratory muscle strength, exercise capacity, physical activity; secondary outcomes are pulmonary functions, peripheral muscle strength, cough strength, respiratory muscle endurance, activity dyspnea perception, quality of life and depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed primary ciliary dyskinesia patients,
* 6-18 years of age,
* under standard medications,
* stable patients without exacerbation or infection

Exclusion Criteria:

* having cognitive disorder,
* orthopedic or neurological disease with a potential to affect functional capacity,
* acute infections or pneumonia,
* problems which may prevent evaluating such as visual problems

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Out- patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | first day
  Evaluated using mouth pressure device
Functional exercise capacity | first day
  Evaluated using 6-minute walking test
Anaerobic exercise capacity | first day
  Evaluated using 3-minute step test
Physical activity | first day
  Evaluated using a metabolic holter

SECONDARY OUTCOMES:
Pulmonary functions | first day
  Evaluated using spirometer
Muscle strength | second day
  Evaluated using hand-held dynamometer for peripheral muscles (shoulder abduction, elbow flexion, knee extension, hand grip strength)
Cough strength | second day
  Evaluated using PEFmeter
Respiratory muscle endurance | second day]
  Evaluated using respiratory muscle trainer (POWERbreathe)
Activity dyspnea | first day
  Evaluated using Modified Borg Scale (0-10 scores, higher values represent a worse outcome)
Generic Quality of life | second day
  Cystic Fibrosis Questionnaire Revised (CFQ-R) Turkish version (Scores range from 0 to 100, with higher scores indicating better health. 9 Quality of life domains:
  Physical, role/school, vitality, emotion, social, body image, eating, treatment burden, health perceptions.3 symptom scales:
  Weight, respiratory, and digestion.Number of items in CFQ-R CFQ-R Teen/Adult: 50. CFQ-R Parent: 44. CFQ-R Child: 35.)
Disease- specific quality of life | second day
  Health-related quality-of-life questionnaires-Primary Ciliary Dyskinesia ( PCD-QOL) Turkish version ( PCD-QOL questionnaire developed different domains for different age groups: pediatric, adolescent, and adult patients as well as parents. These domains mainly evaluate physical, emotional, and social aspects of PCD related to QOL. Moreover, there are different domains for various symptoms at different age groups. The total numbers of items in the questionnaires are 37 in the questionnaire for children, 43 in the one for adolescents, 49 in the one for adults, 41 in the parents' questionnaire.
Depression | second day
  Children's Depression Inventory Turkish Version (Children's Depression Inventory is a 27-item, self-rated, symptom-oriented scale.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Fırat, Pt, Study Chair — Research assistant; Meral Boşnak Güçlü, Pt,Phd, Study Director — Associate professor; Tuğba Şişmanlar Eyüboğlu, MD, Principal Investigator — Medical doctor; Ayşe Tana Aslan, MD,Phd, Principal Investigator — Professor
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Derived] Firat M, Bosnak-Guclu M, Sismanlar-Eyuboglu T, Aslan AT. Aerobic exercise capacity, cough strength, posture, and depression in primary ciliary dyskinesia. Pediatr Pulmonol. 2023 Jan;58(1):73-80. doi: 10.1002/ppul.26158. Epub 2022 Sep 28. PMID 36114723
- [Derived] Firat M, Bosnak-Guclu M, Sismanlar-Eyuboglu T, Tana-Aslan A. Respiratory muscle strength, exercise capacity and physical activity in patients with primary ciliary dyskinesia: A cross-sectional study. Respir Med. 2022 Jan;191:106719. doi: 10.1016/j.rmed.2021.106719. Epub 2021 Dec 17. PMID 34952415
- See also: Related Info — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0071409
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4522020/